CLINICAL TRIAL: NCT01138072
Title: A Phase I, Single-center, Drug Interaction Study Between Simvastatin, Atorvastatin, Rosuvastatin, and GSK2248761 in Healthy Subjects.
Brief Title: A Drug Interaction Study Between Simvastatin, Atorvastatin, Rosuvastatin, and GSK2248761 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 113818
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK2248761, atorvastatin, rosuvastatin, simvastatin, drug interaction, pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — IDX 899; Simvastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Treatment A (Experimental): Simvastatin 20mg (single dose) Day 1
  Interventions: Drug: Simvastatin
- Treatment B (Experimental): Atorvastain 20 mg (single dose) Day 3
  Interventions: Drug: Atorvastatin
- Treatment C (Experimental): Rosuvastatin 10mg (single dose) Day 7
  Interventions: Drug: Rosuvastatin
- Treatment X (Experimental): GSK2248761 200mg single dose Day 10-14, Day 16-17, Day 19-21, Day 23-24
  Interventions: Drug: GSK2248761
- Treatment D (Experimental): GSK2248761 200mg + simvastatin 20 mg Day 15
  Interventions: Drug: GSK2248761; Drug: Simvastatin
- Treatment E (Experimental): GSK2248761 200mg + atorvastatin 20 mg Day 18
  Interventions: Drug: GSK2248761; Drug: Atorvastatin
- Treatment F (Experimental): GSK2248761 200mg + rosuvastatin 20 mg Day 22
  Interventions: Drug: GSK2248761; Drug: Rosuvastatin

INTERVENTIONS:
Drug: GSK2248761 — 200mg once daily
  Arms: Treatment D; Treatment E; Treatment F; Treatment X
Drug: Simvastatin — 20 mg Simvastatin single dose
  Arms: Treatment A; Treatment D
Drug: Atorvastatin — 20 mg atorvastatin single dose
  Arms: Treatment B; Treatment E
Drug: Rosuvastatin — 10 mg rosuvastatin single dose
  Arms: Treatment C; Treatment F

SUMMARY:
This study is a Phase I, open-label, single-sequence drug interaction study to evaluate the effect of repeated doses of GSK2248761 on the pharmacokinetics of simvastatin, atorvastatin, and rosuvastatin in healthy adult subjects. In this study, approximately 14 subjects will receive single doses of simvastatin, atorvastatin, and rosuvastatin on two occasions, once alone and once following administration of repeated doses of GSK2248761. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECGs.
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who: Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 MlU/ml is confirmatory.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Note: this does not include plasma donation.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90 mmHg or heart rate is outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects at Screening and predose Day 1.
* Cardiac conduction abnormalities denoted by any of the following on a single 12-lead ECG at screening or predose Day 1 (a single repeat is allowed for eligibility determination). Including evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome). Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Plasma simvastatin and simvastatin acid Cmax, AUC(0-infinity) and AUC(0-t) following oral administration of a single dose of simvastatin 20mg alone and in combination with GSK2248761 200mg once daily. | 18 days
Plasma atorvastatin Cmax, AUC(0-infinity) and AUC(0-t) following oral administration of a single dose of atorvastatin 20mg alone and in combination with GSK2248761 200mg once daily. | 21 days
Plasma rosuvastatin Cmax, AUC(0-∞) and AUC(0-t) following oral administration of a single dose of rosuvastatin 10mg alone and in combination with GSK2248761 200mg once daily. | 25 days

SECONDARY OUTCOMES:
Plasma ortho and para-hydroxy atorvastatin Cmax, AUC(0-infinity) and AUC(0-t) following oral administration of a single dose of atorvastatin 20mg alone and in combination with GSK2248761 200mg once daily. | 21 days
Plasma simvastatin, simvastatin acid, atorvastatin, ortho and para-hydroxy atorvastatin, and rosuvastatin tmax, t1/2, and percent AUCex. | 25 days
Safety and tolerability parameters including adverse event, concurrent medication, clinical laboratory, ECG, and vital sign assessments. | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Derived] Piscitelli S, Kim J, Gould E, Lou Y, White S, de Serres M, Johnson M, Zhou XJ, Pietropaolo K, Mayers D. Drug interaction profile for GSK2248761, a next generation non-nucleoside reverse transcriptase inhibitor. Br J Clin Pharmacol. 2012 Aug;74(2):336-45. doi: 10.1111/j.1365-2125.2012.04194.x. PMID 22288567